CLINICAL TRIAL: NCT03559959
Title: A Field Experiment to Assess the Demand for HIV Self-Tests in Zimbabwe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Centre for Sexual Health and HIV/AIDS Research Zimbabwe (Other)
Responsible Party: Principal Investigator, Harsha Thirumurthy, Professor, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: MRCZ/A/2199
Record Dates: First submitted 2018-06-05; First posted 2018-06-18 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- $0 price (Experimental): Vouchers for HIV self-testing kits: Individuals will receive a voucher that can be used to redeem an HIV self-testing kit free of charge.
  Interventions: Behavioral: Vouchers for HIV self-testing kits
- $0.5 price (Experimental): Vouchers for HIV self-testing kits: Individuals will receive a voucher that can be used to purchase an HIV self-testing kit at the price of $0.5.
  Interventions: Behavioral: Vouchers for HIV self-testing kits
- $1 price (Experimental): Vouchers for HIV self-testing kits: Individuals will receive a voucher that can be used to purchase an HIV self-testing kit at the price of $1.
  Interventions: Behavioral: Vouchers for HIV self-testing kits
- $2 price (Experimental): Vouchers for HIV self-testing kits: Individuals will receive a voucher that can be used to purchase an HIV self-testing kit at the price of $2.
  Interventions: Behavioral: Vouchers for HIV self-testing kits
- $3 price (Experimental): Vouchers for HIV self-testing kits: Individuals will receive a voucher that can be used to purchase an HIV self-testing kit at the price of $3.
  Interventions: Behavioral: Vouchers for HIV self-testing kits

INTERVENTIONS:
Behavioral: Vouchers for HIV self-testing kits — Participants will be given one referral voucher that offers a self-test kit at a randomly selected price point and distribution site. The vouchers will be valid for one month after the enrollment date. The other household members above 16 years of age will also be offered one voucher per person. Vouchers for the same household will have the same price, distributor, and promotion messages.

SUMMARY:
This study is a field experiment in peri-urban and rural communities near Harare, Zimbabwe, that seeks to estimate the likelihood that individuals will purchase HIV self-tests under various pricing and distribution strategies. About 4,000 adults will be randomly selected, administered a short questionnaire, and given vouchers that will offer them HIV self-tests at randomly allocated prices and distribution sites. The study will also test whether the provision of HIV self-tests can be targeted more cost-effectively to reach high-risk persons and non- recent testers. Last, the study will explore whether demand for repeated HIV self-testing is contingent on the price offered initially.

DETAILED DESCRIPTION:
This study is a field experiment that seeks to obtain "revealed preference" estimates of the likelihood that individuals will purchase oral fluid-based HIV self-tests at alternative prices. Such an approach is useful for estimating the price sensitivity (or elasticity) of demand for HIV self-tests. The study will also estimate the extent to which demand for self-tests differs by certain distribution channels such as retail outlets, public sector health facilities, and other community-based venues. Importantly, the experiment will also test whether the provision of HIV self-tests can be targeted more cost-effectively to reach high-risk persons and non-recent testers by examining the demand for self-tests in these populations in responses to various prices and distribution strategies. The results of the study will provide vital information required by policy makers and implementers on the optical pricing and distribution strategies for introducing HIV self-tests and scaling up HIVST in resource-limited settings. In a subsequent study with additional funding, the study will also seek to determine the long-term implications of offering self-tests at very low prices initially; specifically, it will assess whether free distribution initially suppresses individuals' willingness to pay for self-tests in the future. Roughly 12 months after the initial voucher offer, participants who provided a mobile phone number they can access within their household will be contacted via phone-based text messages and offered the same HIV self-tests again at one common non-zero price. The purchases at 12 months will once again be monitored and linked to participants via a unique identifier that is included in the text messages.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older
* Willing and able to provide written informed consent for participation
* Intends to stay in the study area for at least 12 months

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Voucher redemption | One month after enrollment
  Proportion of individuals that obtained or purchased an HIV self-test

SECONDARY OUTCOMES:
Voucher redemption in key populations | One month
  Proportion of individuals that obtained or purchased an HIV self-test in key segments of the populations, including individuals who have never tested for HIV in the past or not tested recently, individuals with high risk of HIV infection based on self-reported sexual behavior, and individuals with low and high income.

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Thirumurthy, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Zimbabwe and the Centre for Sexual Health and HIV/AIDS Research (CeSHHAR) Zimbabwe, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang W, Matambanadzo P, Takaruza A, Hatzold K, Cowan FM, Sibanda E, Thirumurthy H. Effect of Prices, Distribution Strategies, and Marketing on Demand for HIV Self-testing in Zimbabwe: A Randomized Clinical Trial. JAMA Netw Open. 2019 Aug 2;2(8):e199818. doi: 10.1001/jamanetworkopen.2019.9818. PMID 31461146